CLINICAL TRIAL: NCT02253784
Title: Comparison Between Perineural and Systemic Effect of Dexamethasone as an Adjuvant for Prolongation of Four Nerve Blocks With Bupivacaine in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 14-XX-HYMC
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2014-10

CONDITIONS: Analgesia; Pain, Postoperative
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Dexamethasone; Bupivacaine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group I (ISB-P) (Active Comparator): Four nerve blocks with perineural injection of dexamethasone 0.1 mg/kg and bupivacaine 0.5% - 45 ml
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine
- Group II (ISB-S) (Active Comparator): Four nerve blocks with systemic injection of dexamethasone 0.1 mg/kg and bupivacaine 0.5% - 45 ml
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine
- Group III (ISB-C) (Active Comparator): Four nerve blocks without dexamethasone
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexamethasone
  Arms: Group I (ISB-P); Group II (ISB-S)
Drug: Bupivacaine

SUMMARY:
The addition of dexamethasone (DxaM) to local anesthetic may significantly prolong the duration of a block in total knee arthroplasty. The aim of this study is to determine whether this is a systemic or local effect.

ELIGIBILITY:
Inclusion Criteria:

* Pre-surgical total knee arthroplasty patients

Exclusion Criteria:

* Skin infection near block site
* Allergy to local anesthetics
* Peripheral neuropathy
* Proven opioid dependency
* Coagulopathy
* Dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-10; Primary Completion 2016-10 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Efficacy Perineural DxaM | One day
  Duration of motor and sensory block

SECONDARY OUTCOMES:
Efficacy of Systemic DxaM | One day
  Duration of motor and sensory block

CONTACTS AND LOCATIONS:
Overall Officials: Anatoly Stav, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel